CLINICAL TRIAL: NCT00211211
Title: An International Multicentric, Multidisciplinary Prospective and Randomized Study to Compare Minimally Invasive Reduction and Fixation Using the KyphX System and Radiopaque PMMA Cement to Medical Therapy Alone for the Treatment of Painful, Acute Osteopenic Vertebral Body Compression Fractures
Brief Title: FREE Study - Fracture Reduction Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SP0201 - FREE Study
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2012-01

CONDITIONS: Osteopenia; Osteoporosis; Multiple Myeloma; Bone Neoplasms
Keywords: Osteopenia; Osteoporosis; Multiple Myeloma; Osteolytic Metastatic Tumors; Vertebral Compression Fracture; Back Pain; Spine
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Multiple Myeloma; Bone Neoplasms; Back Pain | interventions — Kyphoplasty

INTERVENTIONS:
Device: Balloon Kyphoplasty

SUMMARY:
The primary objective of this study is to compare the effectiveness of standard medical therapy alone to kyphoplasty using the KyphX system for the treatment of acute vertebral body compression fractures.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of one painful, acute (edema present on MRI obtained within a two weeks period prior to enrolment) thoracic or lumbar (T5-L5) vertebral body compression fracture, due to osteopenia arising from primary or secondary osteoporosis, multiple myeloma, or osteolytic metastatic tumors and maximum of three painful fractures requiring treatment. (NOTE: a T2-weighted MRI should be done unless it is not available);
* Minimum of one acute fracture to be treated that has height loss > 15% of predicted height (average height of two adjacent "normal" vertebrae) when measured at the middle of the vertebral endplate. (NOTE: If the adjacent vertebrae are not normal, the predicted height will be based on the height listed for the fractured vertebra in the table taken from Black et al.)
* Pre-treatment VAS score > 4 on a scale of 10 where 0 is no pain, 5 is moderate pain and 10 is pain "as bad as you can imagine";
* Patient 21 years of age or older;
* The investigator and surgeon/radiologist agree before randomization that the fracture(s) can technically be reduced using an inflatable bone tamp (IBT); and
* A signed Informed Consent is obtained from the patient.

Exclusion Criteria:

* Previous vertebroplasty;
* Vertebral body fracture morphology prevents use of devices (such as endplate below pedicles);
* Pedicle fractures;
* Acute fracture(s) to be treated symptomatic > 3 months at enrollment;
* Pre-existing (not the result of the index fracture) neurological deficit or radicular pain that is not well defined or unstable;
* Spinal cord compression or canal compromise requiring decompression;
* Disabling back pain secondary to causes other than acute fracture;
* Vertebral fracture due to primary or osteoblastic tumors;
* Patient is currently on anticoagulation therapy that can not be interrupted;
* Pre-existing conditions contrary to the kyphoplasty procedure:

  * Systemic infection
  * Local fractured vertebral body infection
  * Temporarily non-reversible bleeding disorder
* Known allergy to any of the drugs, bone void filler material or contrast medium used in the treatment of study subjects
* Dementia and/or inability to give informed consent;
* Inability to walk or stand prior to the vertebral body fracture (walking aids are allowed);
* MRI contraindication (e.g. cerebral aneurysm clips, pacemaker, implanted biostimulators, cochlear implants, penile prosthesis);
* Pregnancy
* Participation in any other clinical trial within the last 30 days.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the effectiveness of standard medical therapy alone to kyphoplasty using the KyphX system for the treatment of acute vertebral compression fractures (VCFs).
Safety will be compared between the study groups throughout the study with focus on clinically meaningful events and subsequent VCFs including the "treated" vertebrae.
The primary study endpoint is the change in quality of life as measured by the Physical Component Summary (PCS) scale of the 36-Item Short Form (SF-36) as measured at the one-month follow-up visit.

SECONDARY OUTCOMES:
The secondary study endpoints are: EuroQol self-report (EQ-5D) questionnaire and SF-36 scores at 1, 3, 6, 12 and 24 months
procedural safety (peri-operative clinical events)
function as measured by objective functionality tests-reaching, "get up and go" and by the subjective Roland Morris disability questionnaire at 1, 3, 6, 12 and 24 months
pain using a 10-point visual analogue scale (VAS) at 5-10 days (post enrollment for the control group and post kyphoplasty for the kyphoplasty group)
changes in spinal deformity as measured radiographically at baseline, 3, 12 and 24 months.
Maintenance of vertebral body height will be assessed from lateral spine x-rays obtained in Kyphoplasty treated subjects only at baseline and at 3, 12, and 24 month visits.
patient satisfaction at 1, 3, 6, 12, 24 months
outcome (nursing home, back to status prior to fracture) at 1, 3, 6, 12, 24 months
economic aspects (including hospital days, disabilities, etc.) at 1, 3, 6, 12, 24 months
the cost-effectiveness of kyphoplasty expressed in incremental cost/quality adjusted life year gained at different time points (1 year and 2 years)
rate of incident fractures at 3, 12 and 24 months (frequency, timing and location)
Each endpoint will be compared between the 2 groups and for its evolution over time.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Johnell, MD, Principal Investigator — UMRA - Malmo, Sweden
Locations (1):
- University of Alabama, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Van Meirhaeghe J, Bastian L, Boonen S, Ranstam J, Tillman JB, Wardlaw D; FREE investigators. A randomized trial of balloon kyphoplasty and nonsurgical management for treating acute vertebral compression fractures: vertebral body kyphosis correction and surgical parameters. Spine (Phila Pa 1976). 2013 May 20;38(12):971-83. doi: 10.1097/BRS.0b013e31828e8e22. PMID 23446769
- [Derived] Ranstam J, Turkiewicz A, Boonen S, Van Meirhaeghe J, Bastian L, Wardlaw D. Alternative analyses for handling incomplete follow-up in the intention-to-treat analysis: the randomized controlled trial of balloon kyphoplasty versus non-surgical care for vertebral compression fracture (FREE). BMC Med Res Methodol. 2012 Mar 24;12:35. doi: 10.1186/1471-2288-12-35. PMID 22443312
- [Derived] Fritzell P, Ohlin A, Borgstrom F. Cost-effectiveness of balloon kyphoplasty versus standard medical treatment in patients with osteoporotic vertebral compression fracture: a Swedish multicenter randomized controlled trial with 2-year follow-up. Spine (Phila Pa 1976). 2011 Dec 15;36(26):2243-51. doi: 10.1097/BRS.0b013e3182322d0f. PMID 21912321
- [Derived] Wardlaw D, Cummings SR, Van Meirhaeghe J, Bastian L, Tillman JB, Ranstam J, Eastell R, Shabe P, Talmadge K, Boonen S. Efficacy and safety of balloon kyphoplasty compared with non-surgical care for vertebral compression fracture (FREE): a randomised controlled trial. Lancet. 2009 Mar 21;373(9668):1016-24. doi: 10.1016/S0140-6736(09)60010-6. Epub 2009 Feb 24. PMID 19246088